CLINICAL TRIAL: NCT05640856
Title: Evaluation of Relationship Between Oxygen Reserve Index and Difficult Airway With Stop Bang Score
Brief Title: Relationship Between STOP BANG Score and Airway Management
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2020-22/16
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Airway Obstruction; Obstructive Sleep Apnea; Hypoxia
Keywords: Oxygen Reserve Index; STOP BANG Score; Difficult Airway
MeSH Terms: conditions — Airway Obstruction; Sleep Apnea, Obstructive; Hypoxia | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D: STOP BANG Score <3
  Interventions: Procedure: intubation
- Group Y: STOP BANG Score ≥ 3
  Interventions: Procedure: intubation

INTERVENTIONS:
Procedure: intubation — Endotracheal tube placement

SUMMARY:
Nowadays, anesthetists may encounter many patients who are not diagnosed with obstructive sleep apnea syndrome (OSAS) to undergo elective surgery. Recognition of these patients by anesthesiologists and taking necessary precautions will significantly reduce perioperative complications and mortality. STOP-BANG is a questionnaire used to predict high risk of OSAS. The aim of our study is to evaluate the clinical use of the oxygen reserve index as an early warning of possible desaturation in patients with low and high risk of OSAS according to the Stop Bang score.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-III
* Between 18-65 years old
* Volunteered to participate in the study

Exclusion Criteria:

* diagnosed with asthma, COPD, heart failure or coronary artery disease, OSAS
* morbidly obese (BMI>45 kg/m2),
* patients with a history of alcohol or drug addiction
* women in pregnancy or lactation
* allergic to the drugs used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 to be intubated undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Oxygenation | up to intubation
  prediction of desaturation by oxygen reserve index in patients with low and high risk of OSAS

SECONDARY OUTCOMES:
Evaluation of difficult Airway | up to intubation
  using mask-ventilation scale in patients with low and high risk of OSAS

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No